CLINICAL TRIAL: NCT07084168
Title: Multimedia Aid for Genetic Testing in Gynecologic Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2417
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Ovary Cancer; Endometrial Cancer
Keywords: genetic testing; video implementation; chart review
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic Testing Awarness (Experimental): Educational videos about genetic testing will be provided for ovarian cancer and endometrial cancer.
  Interventions: Behavioral: Educational videos; Behavioral: Survey

INTERVENTIONS:
Behavioral: Educational videos — Educational videos about genetic testing will be provided. Subjects will be asked to view one of three videos (an endometrial cancer/Lynch Syndrome video or a longer or shorter version of an ovarian cancer video) relevant to their cancer diagnosis and genetic testing.
  Other Names: Genetic testing information
Behavioral: Survey — Subjects will be asked to complete a brief satisfaction survey.

SUMMARY:
This pilot study aims to estimate rates of genetic testing in patients with ovarian and endometrial cancer before and after the implementation of educational videos about genetic testing. Subjects will be asked to view one of three videos relevant to their cancer diagnosis and genetic testing, and have the option to complete a brief satisfaction survey. A chart review to evaluate rates of genetic testing ordered and referrals placed to Genetics before and after the implementation of the videos will be conducted.

Up to 15-20% of ovarian cancer and 3-5% of endometrial cancer is due to inherited genetic mutation. Given this association, the National Comprehensive Cancer Network (NCCN) recommends genetic counseling and testing for all individuals with a diagnosis of ovarian cancer and endometrial cancer. Some challenges to obtaining genetic counseling and testing include missed identification and referral of eligible patients by providers, lack of provider knowledge, and busy clinic visits limiting time for informed consent and maintaining patient autonomy for genetic testing. Although heterogeneous, the literature supports multimedia use in cancer genetics. However, there is a paucity of data in the field of gynecologic oncology for the role of integrating a multimedia approach to genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

* Reviewed informed consent to participate in the study.
* Subject is willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* Diagnosis of ovarian cancer or endometrial cancer
* Eligible for genetic testing
* English or Spanish is the primary language

Exclusion Criteria:

* Previously completed genetic testing
* Did not receive initial cancer-directed treatment at study site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of genetic testing | Baseline
  Proportion of eligible patients undergoing any genetic testing before and after the implementation of educational videos.

SECONDARY OUTCOMES:
Overall rates of genetic testing | Baseline
  Overall rates of genetic testing before and after the implementation of multimedia videos for patient education.
Patient satisfaction | Baseline
  Total scores on patient satisfaction will be measured by a survey. Items are rated by patients on a Likert scale from 1 to 5. Higher scores represent better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tucker, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials